CLINICAL TRIAL: NCT02229474
Title: Identification and Intervention for Dementia in Elderly Africans (IDEA) Study: CST Trial
Brief Title: IDEA Study Cognitive Stimulation Therapy (CST) Trial in Tanzania
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Keith Gray (Other)
Collaborators: Grand Challenges Canada (Other); University of Ibadan (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other); Newcastle University (Other); Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, William Keith Gray, Dr William Gray, Northumbria Healthcare NHS Foundation Trust
Organization: Northumbria Healthcare NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IDEA_TANZANIA_CST1
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-09

CONDITIONS: Dementia
Keywords: Dementia; Cognitive Stimulation Therapy; Quality of life; Cognitive impairment; Africa; Tanzania; Nigeria; Low- and Middle-income countries; Non-pharmacological intervention; Task-shifting; Cognitive screening
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CST intervention (Experimental): We will use a two-group stepped-wedge design. Group 1 will receive the intervention immediately. This will also allow group 2 to act as controls for group 1 and allow further analysis as a controlled trial, during secondary analysis.
  In accordance with the CST manual protocol, patients will be allocated to groups to ensure a spread of abilities and ensure inclusivity. No group contains only one individual of a particular religion or gender, such that they may feel left out. We will allocate patients to groups to avoid excessive travel to the group meeting place, participants may be allocated to a group based on their geographical location.
  Interventions: Behavioral: CST Intervention
- Group 2 (No Intervention): and group 2 will have their intervention delayed until after the end of the group 1 intervention. This will also allow group 2 to act as controls for group 1 and allow further analysis as a controlled trial, during secondary analysis.

INTERVENTIONS:
Behavioral: CST Intervention — The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve quality of life. Sessions will be led and facilitated by a study nurse or occupational therapist. The sessions will be held at a local health centre of village hall.
  Arms: CST intervention

SUMMARY:
This trials of cognitive stimulation therapy (CST) in Tanzania is part of the larger Identification and Intervention for Dementia in Elderly Africans (IDEA) study.

The overall aim of the IDEA study is to set up and evaluate sustainable programmes to facilitate diagnosis of, and therapy for, people with dementia led by local communities in sub-Saharan Africa. We aim seek to improve quality of life for people with dementia and their caregivers.

Within this trial of CST, we hypothesise that CST can significantly improve the quality of people with dementia and their carers living in Africa

DETAILED DESCRIPTION:
Our project will address three specific challenges: 1) Integrate screening and core packages of services into routine primary health care. 2) Provide effective and affordable community-based care and rehabilitation. 3) Develop effective treatment for use by non-specialists, including lay healthcare workers with minimal training.

Dementia is under-diagnosed in sub-Saharan Africa (SSA) and treatment is rarely accessed or available. The burden of dementia on caregivers is high, with loss of income, and psychosocial stress common. However, large scale screening for dementia in such a setting is neither affordable nor sustainable. The purpose of this 3 year project is to provide a sustainable mechanism for diagnosis and therapeutic intervention for people with dementia. We will use 2 complimentary, rural study sites, 1 in Nigeria, West Africa and 2 in Tanzania, East Africa. As a consequence our results should be generalizable to all SSA. Our approach is inexpensive and will have applicability to other low- and middle-income countries.

During Phase I we will validate a screening tool, previously developed by members of our study team from data collected in Tanzania, and carry out a pilot study of the benefits of cognitive stimulation therapy (CST) when used in SSA for those already identified with dementia. During both of these activities we will initiate training of local healthcare workers in diagnosis and management of people with dementia. In Phase II we will engage with local communities to raise awareness of dementia. Building on previous work at both study sites, we will initiate poster, newspaper and radio advertising and use mobile phone text messaging services (for relevant healthcare personnel) to increase awareness of the need to diagnose and intervene at an early stage. We will empower local private pharmacies to help identify people with dementia, a relationship which will ultimately be mutually beneficial through the supply of medicines to treat risk factors for dementia, such as hypertension. We will engage with local community leaders and government officials to assist us in this awareness raising, an approach that has proven successful in previous studies by our team in SSA. One of our study team (Dr Mushi (DM)) is a social scientist based in Tanzania and during Phase II we will conduct qualitative research into attitudes and beliefs surrounding dementia and identify any barriers to diagnosis in both sites. The results of this research will be fed back to inform other phases of the study. Finally, in phase III we will initiate a program of community based CST led by local occupational therapists (OTs) and nurse specialists. OTs and nurses will train caregivers in CST techniques and we hope that the training will ultimately be led by caregivers allowing such therapy to become sustainable within communities in the longer term. We will evaluate changes in cognition in people with dementia, and quality of life (QOL) in both people with dementia and their caregivers, post-intervention. We will carry out a full economic evaluation of the effect of our program, to be led by a heath economist based at Newcastle University, United Kingdom.

This protocol cover the CST trial (Phase III of the study) in Tanzania

ELIGIBILITY:
Inclusion Criteria:

* Anyone with dementia living within the study site

Exclusion Criteria:

* The participant and the family should have consented to take part in the study.
* Unable to travel to the centre where the CST sessions will be held due to physical impairment (e.g. bedbound or immobile)
* After assessment by the study doctor, deemed unable to engage in CST sessions (e.g. follow instructions and participate in activities) due to severe physical or cognitive impairment.
* Profound deafness
* Total blindness
* Aphasia - they should be able to understand verbal communication and communicate verbally (mild impairments are acceptable).
* The participant should be able to sit in a group setting for 1 hour.
* There should not be agitation, depression or psychosis to an extent that the person would not be able to tolerate spending time with other people in a group setting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adesola Ogunniyi, MD, Principal Investigator — University of Ibadan, Ibadan, Nigeria; Richard W Walker, MD, Study Chair — Northumbra Healthcare NHS Foundation Trust; Delare Mushi, Study Director — Kilimanjaro Christian Medical University College; Catherine L Dotchin, MD, Study Director — Northumbria Healthcare NHS Foundation Trust; William K Gray, PhD, Study Director — Northumbria Healthcare NHS Foundaion Trust
Locations (1):
- Hai district DSS, Moshi, Kilimanjaro, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
We will publish our findings in academic journals and state that we will make anonymized participant level data available in the manuscript, upon request to the authors.

REFERENCES:
- [Background] Longdon AR, Paddick SM, Kisoli A, Dotchin C, Gray WK, Dewhurst F, Chaote P, Teodorczuk A, Dewhurst M, Jusabani AM, Walker R. The prevalence of dementia in rural Tanzania: a cross-sectional community-based study. Int J Geriatr Psychiatry. 2013 Jul;28(7):728-37. doi: 10.1002/gps.3880. Epub 2012 Sep 20. PMID 22996739
- [Background] Gray WK, Paddick SM, Kisoli A, Dotchin CL, Longdon AR, Chaote P, Samuel M, Jusabani AM, Walker RW. Development and Validation of the Identification and Intervention for Dementia in Elderly Africans (IDEA) Study Dementia Screening Instrument. J Geriatr Psychiatry Neurol. 2014 Jun;27(2):110-8. doi: 10.1177/0891988714522695. Epub 2014 Feb 26. PMID 24578459
- [Derived] Lok N, Buldukoglu K, Barcin E. Effects of the cognitive stimulation therapy based on Roy's adaptation model on Alzheimer's patients' cognitive functions, coping-adaptation skills, and quality of life: A randomized controlled trial. Perspect Psychiatr Care. 2020 Jul;56(3):581-592. doi: 10.1111/ppc.12472. Epub 2020 Jan 12. PMID 31930518

RESULTS

PARTICIPANT FLOW:
Groups:
- CST Intervention: We will use a two-group stepped-wedge design. Group 1 will receive the intervention immediately. This will also allow group 2 to act as controls for group 1 and allow further analysis as a controlled trial, during secondary analysis.
  CST Intervention: The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve quality of life. Sessions will be led and facilitated by a study nurse or occupational therapist. The sessions will be held at a local health centre of village hall.
Period: Overall Study
Arm/Group | CST Intervention | Group 2
Started | 16 | 18
Completed | 16 | 15
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- CST Intervention: We will use a two-group stepped-wedge design. Group 1 will receive the intervention immediately. This will also allow group 2 to act as controls for group 1 and allow further analysis as a controlled trial, during secondary analysis.
  In accordance with the CST manual protocol, patients will be allocated to groups to ensure a spread of abilities and ensure inclusivity. No group contains only one individual of a particular religion or gender, such that they may feel left out. We will allocate patients to groups to avoid excessive travel to the group meeting place, participants may be allocated to a group based on their geographical location.
  CST Intervention: The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve outcomes
- Total: Total of all reporting groups
Arm/Group | CST Intervention | Group 2 | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 81 [76 to 86] | 80 [74 to 86] | 80 [76 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization Brief Quality of Life Scale
Description: The WHOQOL-Bref will assess quality of life in patients and carers. The scale is scored from a minimum of 4 to a maximum of 20, with higher scores indicating better quality of life. The scores are measured as units on a scale
Time Frame: Baseline
Population: Analysis for QOL data comparing pre- and post intervention scores
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- CST Intervention: We will use a two-group stepped-wedge design. Group 1 will receive the intervention immediately. This will also allow group 2 to act as controls for group 1 and allow further analysis as a controlled trial, during secondary analysis.
  In accordance with the CST manual protocol, patients will be allocated to groups to ensure a spread of abilities and ensure inclusivity. No group contains only one individual of a particular religion or gender, such that they may feel left out. We will allocate patients to groups to avoid excessive travel to the group meeting place, participants may be allocated to a group based on their geographical location.
  CST Intervention: The CST intervention comprises 14 sessions lasting 1-2 hours across 7 weeks. The CST manual has been adapted for use in this setting by members of our study team. Each session has a theme. Activities include tasks aimed at engaging participants in cognitive and physical tasks designed to improve quality of life.
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 2.5 [2 to 3] | 2 [1 to 4]

2. Primary Outcome: World Health Organization Brief Quality of Life Scale
Description: The WHOQOL-Bref will assess quality of life in patients and carers. The WHOQOL-Bref will assess quality of life in patients and carers. The scale is scored from a minimum of 4 to a maximum of 20, with higher scores indicating better quality of life. The scores are measured as units on a scale
Time Frame: Immediately post-intervention
Population: Groups attending CST sessions
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 2.5 [1 to 4] | 2.5 [1 to 4]

3. Secondary Outcome: World Health Organization Brief Quality of Life Scale
Description: The scale will assess quality of life in patients and carers. The scale is scored from a minimum of 4 to a maximum of 20, with higher scores indicating better quality of life. The scores are measured as units on a scale.
Time Frame: Four weeks post intervention
Population: people atending CST sessions
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 2.5 [1 to 4] | 2.5 [1 to 4]

4. Secondary Outcome: Identification and Intervention for Elderly Africans Cognitive Screen
Description: The screen will assess cognitive function. It is scored from a minimum of 0 to a maximum of 15, with a higher score indicating better cognitive function.
Time Frame: Baseline
Population: people attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 6 [4.25 to 8] | 5 [3.75 to 8]

5. Secondary Outcome: Adapted Alzheimer's Disease Assessment Scale-cognitive Scale
Description: The adapted scale will assess cognitive function, specifically change in function over time. The minimum possible score is 0 and the maximum is 69. A lower score indicates better cognitive function.
Time Frame: Baseline
Population: people attending CST
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 31.5 (8.358) | 27.4 (6.647)

6. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: The scale will assess anxiety and depression in patients and carers. The maximum possible score is 21 and the minimum score is 0. Lower score indicates lower levels of anxiety and depression.
Time Frame: Baseline
Population: People attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 8 [4.5 to 12.75] | 5.5 [3.75 to 11.25]

7. Secondary Outcome: Zarit Burden Interview
Description: The scale will assess carer burden. There are 22 questions each scored from 0 to 4. Overall, the scale is scored from 0 to 88, with a higher score indicating greater burden.
Time Frame: Baseline
Population: People attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 12.5 [10.25 to 20.75] | 17.5 [10.75 to 24.0]

8. Secondary Outcome: Identification and Intervention for Elderly Africans Cognitive Screen
Description: as for outcome 4
Time Frame: Immediately post-intervention
Population: People attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 5 [4 to 8] | 6.5 [4.75 to 8.0]

9. Secondary Outcome: Adapted Alzheimer's Disease Assessment Scale-cognitive Scale
Description: as for outcome 5
Time Frame: Immediately post-intervention
Population: People attending CST
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 23.4 (8.560) | 26.6 (7.121)

10. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: as for outcome 6
Time Frame: Immediately post-intervention
Population: People attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 9.0 [8.0 to 13.0] | 7.5 [3.5 to 11.25]

11. Secondary Outcome: Zarit Burden Interview
Description: as for outcome 7
Time Frame: Immediately post-intervention
Population: people attending CST
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CST Intervention | Group 2
Number analyzed (Participants) | 16 | 18
units on a scale | 9.5 [5.75 to 16.75] | 13.0 [9.5 to 22.0]

ADVERSE EVENTS:
Arm/Group | CST Intervention | Group 2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No